CLINICAL TRIAL: NCT06610877
Title: Ultrasound Neuromodulation in Essential Tremor
Acronym: UNMET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Focused Ultrasound Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P0573974
Record Dates: First submitted 2024-09-20; First posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Essential Tremor; Neuromodulation
Keywords: Essential Tremor; Neuromodulation; Focused Ultrasound; brain functional connectivity
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Intervention Model Description: This is a within-subject repeated-measures interventional study to test which of a set of LIFU stimulation parameters are most effective at producing temporary tremor reduction when applied to the DRTT - the white matter circuit involved in essential tremor. During a single session up to 25 different stimulation protocols will be tested in each participant in a shuffled manner including sham stimulation protocols.
Masking Description: Participants will be unaware of which focused ultrasound protocols are being applied when or whether the applied protocol is considered to be a candidate active stimulation or sham protocol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- To determine the most effective stimulation parameters for DRTT LIFU neuromodulation. (Experimental): Investigators will record wrist accelerometer signals while participants maintain standardized postures that maximally elicit their tremor before, during, and after delivering LIFU stimulation.
  Interventions: Device: Focused Ultrasound Neuromodulation

INTERVENTIONS:
Device: Focused Ultrasound Neuromodulation — Each ultrasound stimulation protocol will last for 60 seconds, consisting of 4 pulse trains of 5 seconds duration separated by 10 second intervals without stimulation. Across successive stimulation protocols (up to 25/patient) investigators will systematically vary pulse repetition frequency, duty cycle, and acoustic intensity to determine how these parameters contribute to the behavioral effect (transient tremor reduction). Parameters will be shuffled to control for group-level carry over effects and will include sham (unfocused or off-target stimulation) conditions to control for non-specific auditory confounds.
  Other Names: Sham stimulation with defocused or off-target sonication
Device: Focused ultrasound neuromodulation — Each ultrasound stimulation protocol will last for 60 seconds, consisting of 4 pulse trains of 5 seconds duration separated by 10 second intervals without stimulation. Across successive stimulation protocols (up to 25/patient) investigators will systematically vary pulse repetition frequency, duty cycle, and acoustic intensity to determine how these parameters contribute to the behavioral effect (transient tremor reduction) in each patient. Parameters will be shuffled to control for group-level carry over effects and will include sham (unfocused or off-target stimulation) conditions to control for non-specific auditory confounds.

SUMMARY:
This study is being done to test whether low-intensity focused ultrasound (LIFU) (low energy sound waves) cause temporary changes in brain activity and behavior when directed at particular parts of the brain. By targeting LIFU to the parts of the brain thought to be responsible for essential tremor (ET), and measuring any associated improvement in tremor, the investigators hope to show that LIFU can be a useful tool for studying the brain circuits responsible for tremor and other brain disorders.

DETAILED DESCRIPTION:
Hypothesis

Precisely targeted low-intensity focused ultrasound (LIFU) modulation of the dentatorubrothalamic tract (DRTT) results in transient improvement of essential tremor (ET). DRTT LIFU neuromodulation produces functional connectivity changes that mirror brain network changes after MR-guided high-intensity focused ultrasound (HIFU) thalamotomy.

Aims

1. To determine the optimal stimulation parameters for DRTT LIFU neuromodulation: the investigators will record wrist accelerometer signals while systematically varying pulse repetition frequency, duty cycle, and acoustic intensity.
2. To map network effects of DRTT LIFU neuromodulation: the investigators will record resting state fMRI (rs-fMRI) immediately after DRTT LIFU neuromodulation with the parameters most effective at reducing tremor in each patient.

Design

This is a within-subject repeated-measures interventional study designed to determine the set of LIFU stimulation parameters that are maximally effective at producing a temporary tremor reduction when applied to the DRTT - the white matter circuit in the brain in which abnormal activity causes essential tremor.

The investigators will recruit patients from the established MR-guided high-intensity focused ultrasound (HIFU) ET program at UCSF (which treats 6-9 patients/month). Due to the logistical complexity of performing MRI in patients with MR-conditional pacemakers (need for device and patient monitoring), patients with pacemakers will be excluded from enrollment. Study inclusion criteria will otherwise be similar to those for the HIFU procedure itself, namely medically refractory tremor that is expected to improve with HIFU thalamotomy without contraindications to MRI or inability to stop anticoagulation. As part of their routine pre-procedure evaluation these patients receive a dedicated head CT for calculation of skull density ratio (SDR) and a 3T brain MRI that includes high resolution diffusion imaging for tractography to identify the DRTT, as well as specialized anatomic scans (including proton density (PD) and white matter nulled T1 (wm-null T1) sequences to define adjacent thalamic anatomy.

Study participants will undergo a single LIFU session lasting 3-4 hours, generally in the 1-2 days prior to their HIFU treatment. The investigators will perform LIFU stimulation using a commercially available, portable, neuronavigated focused ultrasound system (NeuroFUS PRO, BrainBox, Cardiff, UK) and will target LIFU stimulation using the same image-guided protocol used for the patient's subsequent HIFU treatment. Wrist-based accelerometers (MP160 + TSD109A; BIOPAC Systems, Inc.) will be used to provide a quantitative behavioral readout of the LIFU effect. The investigators will use power spectrum density analysis of accelerometer signals to quantify the severity of tremor before and after LIFU and HIFU sonications. To evaluate the effect of DRTT LIFU on tremor severity and the contribution of the different acoustic parameters tested, the investigators will perform individual- and group-level statistical analyses on the quantified tremor power in the characteristic ET range of 4-12 Hz. The hair on the participant's head will be shave at the start of the session to facilitate the passage of the ultrasound energy (an existing requirement of the subsequent HIFU treatment).

The transient nature of LIFU tremor reduction (on the order of 10-20 minutes) will facilitate high-throughput parameter screening through repeated sonications within the same session (up to 25, depending on patient response). Stimulation protocols consisting of 5 seconds of active stimulation followed by 10 seconds of no stimulation repeated four times (total 60 s) will be delivered using a range of sample parameters. Stimulation parameters will be shuffled in each session to control for carryover effects at the group level. After each 60-s stimulation, there will be a 3 minute inter-stimulation period, during which tremor severity will be monitored every 60 seconds through quantitative accelerometer recordings. If a change in tremor severity greater than 50% is found in the post-LIFU period compared to the pre-LIFU baseline, the investigators will wait until tremor returns to a level comparable to baseline before proceeding with additional stimulations. A similar approach was followed in a recent study by Aubry et al. (2024) with the Insightec Exablate system. The entire LIFU stimulation session will last approximately 100 minutes, sufficient to screen up to 25 stimulation protocols (1 min sonication + 3 min wait per protocol) depending on tremor response.

At the end of the session, the investigators will identify the stimulation parameters that produced the largest tremor suppression compared to the respective pre-LIFU baseline. They will then deliver a sham (off-target or defocused) sonication using these maximally effective parameters to control for nonspecific sensory and auditory effects evoked by the ultrasound stimulation. Following this, the investigators will perform a final active sonication targeting the DRTT with the maximally effective parameters, this final stimulation will be immediately followed by a brief (~20-30 minute) MRI scan to measure the effects of LIFU on brain functional connectivity derived from rs-fMRI.

Patients will then proceed with their scheduled HIFU treatment, which will include similar intra-procedure wrist-base accelerometer measurements to document behavioral effects of HIFU on ET, as well as post treatment MRI to evaluate for post-treatment complications and to measure the effects of HIFU on brain functional connectivity as assessed with rs-fMRI.

ELIGIBILITY:
Inclusion Criteria:

* Patients with medically refractory tremor scheduled to undergo MR-guided high-intensity focused ultrasound (HIFU) thalamotomy to treat their tremor at UCSF.

Exclusion Criteria:

* Due to the logistical complexity of performing MRI in patients with MR-conditional pacemakers (need for device and patient monitoring), patients with pacemakers will be excluded from enrollment. All other patients undergoing HIFU thalamotomy for tremor will be eligible for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Reduction in tremor tremor | For 3 minutes immediately after the application of each sonication protocol
  The investigators will screen ultrasound parameters through repeated sonications within the same session (up to 25, depending on patient response) to determine which parameter set is most effective at reducing tremor in each participant as measured by wrist accelerometers (reduction in tremor power from baseline in the characteristic ET range of 4-12 Hz). Stimulation protocols will consist of 5 seconds of active stimulation followed by 10 seconds of no stimulation repeated four times (total 60 s). After each 60-s stimulation, there will be a delay of 3 minutes, during which the investigators will monitor tremor severity every 60 seconds through quantitative accelerometer recordings. If a change in tremor severity greater than 50% is found in the post-LIFU period compared to the pre-LIFU baseline, the investigators will wait until tremor returns to a level comparable to baseline before proceeding with additional stimulations.

SECONDARY OUTCOMES:
Changes in functional connectivity of brain networks | 20-30 min MRI scan at the end of the 3-4 hour experimental session
  The investigators will record resting state fMRI (rs-fMRI) immediately after DRTT LIFU neuromodulation with the parameters most effective at reducing tremor in each patient. The investigators hypothesize that LIFU neuromodulation will result in systematic changes in functional connectivity in motor-related brain networks between pre-LIFU (baseline) imaging and immediate post-LIFU imaging. These changes will additionally be compared to those observed between baseline imaging and post-HIFU imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Leo Sugrue, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- Pritzker Building, UCSF, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No